CLINICAL TRIAL: NCT04015817
Title: Impact of an Interdisciplinary Approach in the Management of Refractory Dyspnoea on Patients' Quality of Life by a Respiratory Care Team Non-specialized in Palliative Care
Brief Title: Interdisciplinary Approach for Refractory Dyspnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ligue Pulmonaire Neuchâteloise (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LPNE_02
Record Dates: First submitted 2019-07-01; First posted 2019-07-11 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Dyspnea
Keywords: Dyspnea; Well being; respiratory care team non-specialized in palliative care
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Etude longitudinale (Experimental): Work on positions, ventilatory education, use of a fan, pulmonary rehabilitation, stress management, mindfulness meditation, psychosocial services, support from the mobile palliative care team
  Interventions: Other: paramedical and non-pharmacological services

INTERVENTIONS:
Other: paramedical and non-pharmacological services — Paramedical and non-pharmacological services (work on positions, ventilatory education, use of a fan, pulmonary rehabilitation, stress management, mindfulness meditation, psychosocial services, possible support from the mobile palliative care team)

SUMMARY:
Dyspnoea is a very common symptom in many diseases, not only cardiorespiratory, but also renal or neurological diseases. It can be defined as " difficult, laboured and uncomfortable breathing […]. It is a subjective symptom. As pain, it involves both the patient's perception of the sensation and his reaction to it ". It can occur during even moderate effort and sometimes also at rest and tends to increase as the disease causing it progresses. Dyspnoea has therefore a significant on the various aspects of the patient's daily life and those around him or her (travel, leisure, daily activities, etc.) leading to a decrease in quality of life and possibly to anxiety and/or depressive symptoms. Among a vulnerable, elderly population that benefits from home care, it affects more than 46 % of patients in north-west of Switzerland.

Despite the handicap generated by daily dyspnoea, this complaint is often difficult to recognize by health professionals or family and friends, due in particular to a feeling of helplessness in the care provided. In addition, the treatment of the disease responsible for dyspnoea by the doctor does not always provide relief.

In this context, it is essential that people with dyspnoea, families and friends are supported in their experiences and acquire techniques and alternatives that help them better manage dyspnoea on a daily basis.

The first objective is to evaluate the feasibility of a dyspnoea support program led by a respiratory care team non-specialized in palliative care and its effect on quality of life and control of dyspnoea symptoms by patients .

A second objective is to measure patient's satisfaction about the program.

DETAILED DESCRIPTION:
The dyspnoea support program will include 4 steps:

Step 1: Initial interview Before the initial interview, the responsible physician will review or examine the medical records via the request sheet sent by the referring physician or pneumologist containing the patient's diagnoses, history and medications. These files will then be sent to the team coordinator.

The team coordinator will meet the patient to obtain complete informations about his or her experiences with dyspnoea. Validated written questionnaires in French will be completed to complete the evaluation:

* Edmonton Symptom Assessment scale (ESAS):
* London Chest Activity of Daily Living (LCADL):
* Hospital Anxiety and Depression scale (HADS):
* Chronic Respiratory disease questionnaire (CRQ):

Blood oxygen saturation (Sp02) without O2 will be measured for each patient. If deemed necessary by the responsible physician (Dr. Clark) to complete the evaluation, a spirometry and an Incremental Shuttle Walk Test (ISWT) test will be performed by a physiotherapist.

Step 2: Specialized appointment:

The coordinator will review the patient to present the measures and strategies that will be proposed according to his/her needs and with reference to the evaluation carried out. An anti-dyspnoea checklist providing advice, useful information and exercises to better manage dyspnoea in daily living will be provided, as well as a self-observation logbook to optimize self-energy and fatigue management.

Step 3: Services:

The measures proposed by the coordinator and accepted by the patient will be implemented, for example: work on positions, ventilatory education, use of a fan, pulmonary rehabilitation, stress management, mindfulness meditation, psychosocial services, possible support from the mobile palliative care team, etc. As the measures proposed depend on the evaluation carried out, this is an individualised program. Different measures can be combined in various ways and successions to meet the needs of the patient.

Step 4: Assessment of progress:

Once the program is completed, evolution of dyspnoea perception following the program will be evaluated. CRQ and HADS questionnaires will be completed and patient's satisfaction will be evaluated (look "statistical consideration").

After the program, a follow-up is planned: patients will be seen again at 3 and 6 months after the program. It will then be a matter of completing the CRQ and HADS questionnaires and monitoring the patients' progress.

ELIGIBILITY:
Inclusion Criteria:

* refractory breathlessness on exertion or rest (Medical Research Council (MRC) dyspnea scale score ≥2), despite optimum treatment of the underlying disease, as deemed by the responsible physician;
* advanced disease such as cancer, chronic obstructive pulmonary disease (COPD), chronic heart failure, interstitial lung disease or motor neuron disease;
* willing to engage with proposed therapy (physiotherapy);
* able to provide informed consent in French.

Exclusion Criteria:

* Breathlessness of unknown cause;
* A primary diagnosis of chronic hyperventilation syndrome;
* Completely house (or hospital or nursing home) bound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change measured by the Chronic Respiratory Questionnaire (CRQ) between the initial interview (T0) and the progress report in patients with refractory dyspnea | an average of four month
  Minimally important difference is reflected by a change in score of 0.5 on a 7 point scale

SECONDARY OUTCOMES:
Measure patient satisfaction with the program in the progress report : visual analogic scale | an average of four month
  Satisfaction assessment using a visual analogic scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Fellrath, Prof, Principal Investigator — Hopital Neuchatelois
Locations (1):
- Ligue pulmonaire neuchâteloise, Peseux, Canton of Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the data collected with other researchers.

REFERENCES:
- [Background] Booth S, Burkin J, Moffat C, Spathis A. Managing Breathlessness in Clinical Practice. 1st ed. New York : Springer; 2013. 265 p.
- [Background] Comroe, J. Some theories on the mechanism of dyspnea. In: Howell J, Campbell, E. Breathlessness: proceeding of an international symposium on breathlessness. Oxford: Blackwell; 1965.
- [Background] Higginson IJ, Bausewein C, Reilly CC, Gao W, Gysels M, Dzingina M, McCrone P, Booth S, Jolley CJ, Moxham J. An integrated palliative and respiratory care service for patients with advanced disease and refractory breathlessness: a randomised controlled trial. Lancet Respir Med. 2014 Dec;2(12):979-87. doi: 10.1016/S2213-2600(14)70226-7. Epub 2014 Oct 29. PMID 25465642
- [Background] Clark, G, Marechal, M. COPD knowledge in a swiss frail selected population. European respiratory Society Congress 2018
- [Background] Pautex S, Vayne-Bossert P, Bernard M, Beauverd M, Cantin B, Mazzocato C, Thollet C, Bollondi-Pauly C, Ducloux D, Herrmann F, Escher M. Validation of the French Version of the Edmonton Symptom Assessment System. J Pain Symptom Manage. 2017 Nov;54(5):721-726.e1. doi: 10.1016/j.jpainsymman.2017.07.032. Epub 2017 Jul 25. PMID 28751077
- [Background] Beaumont M, Couturaud F, Jego F, Pichon R, Le Ber C, Peran L, Roge C, Renault D, Narayan S, Reychler G. Validation of the French version of the London Chest Activity of Daily Living scale and the Dyspnea-12 questionnaire. Int J Chron Obstruct Pulmon Dis. 2018 Apr 30;13:1399-1405. doi: 10.2147/COPD.S145048. eCollection 2018. PMID 29750026
- [Background] Bocerean C, Dupret E. A validation study of the Hospital Anxiety and Depression Scale (HADS) in a large sample of French employees. BMC Psychiatry. 2014 Dec 16;14:354. doi: 10.1186/s12888-014-0354-0. PMID 25511175
- [Background] Bourbeau J, Maltais F, Rouleau M, Guimont C. French-Canadian version of the Chronic Respiratory and St George's Respiratory questionnaires: an assessment of their psychometric properties in patients with chronic obstructive pulmonary disease. Can Respir J. 2004 Oct;11(7):480-6. doi: 10.1155/2004/702421. PMID 15505701